CLINICAL TRIAL: NCT03700996
Title: Clinical Outcome Following Arthroscopic Knee Surgery (COFAKS)
Brief Title: Clinical Outcome Following Arthroscopic Knee Surgery
Acronym: (COFAKS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Memorial Hermann Hospital (Other)
Responsible Party: Principal Investigator, Lane Bailey, Director of Research and Education, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MH-14-0734 (Parent Study)
Record Dates: First submitted 2018-09-26; First posted 2018-10-09 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: ACL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: There are no existing data available to guide clinicians in the appropriate rehabilitation progression of patients who have undergone knee arthroscopy. The investigator intends to fill this void by establishing normative recovery curves for patients undergoing knee arthroscopy.

Research Design: Prospective Observational Design Procedures: Patients 10-70 years old will be screened for "standard of care" clinical and functional outcomes to occur at standardized time-points (post-op weeks 1-4, 8, 12, 16, 20 and return to sport/activity) following arthroscopic knee surgery. Recovery curves will be plotted for all outcome variables of interest including; (1) International knee Disability Committee (IKDC) survey, (2) Tampa Kinesiophobia scale, (3) Tegner activity scale, (4) Marx activity scale, (5) Passive knee range of motion/heel-height difference, (6) Balance Error Scoring System (BESS), (7) Quad/Hamstring strength ratios, (8) Y-Balance, (9) Functional Movement Screening, (10) Vail-Sport Test, (11) Landing Error Scoring System (LESS), (12) Hop Testing, and the (13) Sports Metrics Test. Polynomial lines-of-best-fit and 95% confidence intervals will be plotted to provide objective recovery curves for clinical utilization and stratification of patient recovery.

Risks: There are no additional risks to "standard physical therapy practice" for post-surgical patients participating in this study. The investigator will not be using invasive procedures or testing modalities that emit radiation.

Benefits & Clinical Relevance: This information may offer valuable information to clinicians treating patients following knee arthroscopy by providing objective data for each phase of post-operative recovery. Identifying key landmarks and functional milestones may allow the ability to identify patients who are not meeting clinical expectations and subsequently tailor rehabilitation programs to improve recovery trajectories.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10-70; undergoing primary knee arthroscopy; & participating in post-operative physical therapy management.

Exclusion Criteria:

* Patients will be excluded from the study if they elect to not have knee arthroscopy. Have other orthopedic or medical complications (fractures, deep vein thrombosis,) that would be a contraindication to standard post-operative physical therapy care.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Exclusion Criteria:
  * will be surgical candidates who have elected surgical intervention for internal derangement of the knee.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-10-23 (Actual); Primary Completion 2021-12-23 (Estimated); Study Completion 2021-12-23 (Estimated)

PRIMARY OUTCOMES:
International Knee Disability Committee (IKDC) Survey | Post op week 4
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 5
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 6
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 7
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 8
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 9
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 10
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 11
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 12
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 13
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 14
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 15
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 16
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 17
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 18
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 19
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week 20
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
International Knee Disability Committee (IKDC) Survey | Post op week Return to Sport: range 21 weeks to 52 weeks
  Self-Report Outcomes:
  The International Knee Disability Committee Survey is an 18-item instrument designed to measure pain, symptoms, function and sports activity in patients with a variety of knee conditions. A sum score is calculated and then transformed to a 100-point scale, with 100 indicating no restrictions in daily and sports activities and the absence of symptoms. The overall score will be reported.
Marx Scale | Post op week 4
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 5
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 6
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 7
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 8
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 9
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 10
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 11
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 12
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 13
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 14
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 15
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 16
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 17
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 18
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 19
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week 20
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Marx Scale | Post op week Return to Sport: range 21 weeks to 52 weeks
  Self-Report Outcomes:
  MARX focuses on four activity points: running, deceleration, cutting (changes directions while running), and pivoting. The four knee functions are rated on a 5-point scale of frequency and scores added up to a maximum of 16 points with a higher score indicating more frequent participation.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 4
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 5
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 6
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 7
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 8
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 9
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 10
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 11
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 12
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 13
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 14
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 15
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 16
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 17
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 18
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 19
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week 20
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | Post op week Return to Sport: range 21 weeks to 52 weeks
  Self-Report Outcomes:
  Scale consists of 12 questions regarding the psychological impact of returning to sports in the sports population. The items are scored on a visual analogical scale from 0 to 100. With 100 being the better outcome. The overall score will be reported.
Range of Motion | Post op week 4
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 5
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 6
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 7
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 8
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 9
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 10
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 11
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 12
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 13
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 14
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 15
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 16
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 17
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 18
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 19
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week 20
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Range of Motion | Post op week Return to Sport: range 21 weeks to 52 weeks
  Clinical Measures:
  The normal movement of the knee measured in degrees from the center of the knee. The instrument used to take the measurement is called a double-armed goniometer.
Y-Balance | Post op week 8
  Physical Performance
Y-Balance | Post op week 9
  Physical Performance
Y-Balance | Post op week 10
  Physical Performance
Y-Balance | Post op week 11
  Physical Performance
Y-Balance | Post op week 12
  Physical Performance
Y-Balance | Post op week 13
  Physical Performance
Y-Balance | Post op week 14
  Physical Performance
Y-Balance | Post op week 15
  Physical Performance
Y-Balance | Post op week 16
  Physical Performance
Y-Balance | Post op week 17
  Physical Performance
Y-Balance | Post op week 18
  Physical Performance
Y-Balance | Post op week 19
  Physical Performance
Y-Balance | Post op week 20
  Physical Performance
Y-Balance | Post op week Return to Sport: range 21 weeks to 52 weeks
  Physical Performance
Single Leg Hop | Post op week 8
  Physical Performance
Single Leg Hop | Post op week 9
  Physical Performance
Single Leg Hop | Post op week 10
  Physical Performance
Single Leg Hop | Post op week 11
  Physical Performance
Single Leg Hop | Post op week 12
  Physical Performance
Single Leg Hop | Post op week 13
  Physical Performance
Single Leg Hop | Post op week 14
  Physical Performance
Single Leg Hop | Post op week 15
  Physical Performance
Single Leg Hop | Post op week 16
  Physical Performance
Single Leg Hop | Post op week 17
  Physical Performance
Single Leg Hop | Post op week 18
  Physical Performance
Single Leg Hop | Post op week 19
  Physical Performance
Single Leg Hop | Post op week 20
  Physical Performance
Single Leg Hop | Post op week Return to Sport: range 21 weeks to 52 weeks
  Physical Performance

CONTACTS AND LOCATIONS:
Overall Officials: Lane Bailey, Principal Investigator — Memorial Hermann Hospital
Locations (1):
- The University of Texas Health Science Center-Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No